CLINICAL TRIAL: NCT01148160
Title: The Correlation of Voriconazole Trough Plasma Levels With Genetic Polymorphism, Efficacy, and Safety Outcomes in Hematologic Malignancy Patients With Invasive Pulmonary Aspergillosis
Brief Title: Voriconazole Trough Plasma Levels : Genetic Polymorphism, Efficacy, Safety in Patients With Hematologic Malignancy
Status: Terminated | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Assistantant Professor, Asan Medical Center
Other Study IDs: VCZ-IPA-HEM-2010
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Invasive Fungal Infection
Keywords: voriconazole; invasive pulmonary aspergillosis; hematologic malignancy; therapeutic drug monitoring; genetic polymorphism; efficacy; safety
MeSH Terms: conditions — Invasive Fungal Infections; Invasive Pulmonary Aspergillosis; Hematologic Neoplasms | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Venous blood sampling will be carried out at steady state for therapeutic drug monitoring(trough sampling:right before the dose)
  * Genotyping will be performed using peripheral blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with hematologic malignancies who were given voriconazole to treat invasive (pulmonary) aspergillosis at Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
  Interventions: Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — intravenous, oral administration

SUMMARY:
Multiple factors are associated with a large variability in voriconazole exposure following standard dose administration, such as non-linear saturable pharmacokinetics, drug-drug interactions, liver disease, patient age, and genetic polymorphism of the metabolic enzymes.

Voriconazole is extensively metabolized by the human hepatic enzymes, primarily mediated by CYP2C19. The polymorphisms account for a relatively large portion of inter-individual variance observed in voriconazole plasma concentrations.

However, there are limited data on the relationships between voriconazole blood levels and clinical outcomes or safety in Asian populations.

The purpose of this study is to investigate the relationships of voriconazole blood levels with genetic polymorphism, safety, and clinical outcomes in immunocompromised patients with invasive pulmonary aspergillosis.

DETAILED DESCRIPTION:
The investigators are trying to establish that routine clinical practice for voriconazole therapeutic drug monitoring can improve the efficacy and safety outcomes.

In Korean patients with hematologic malignancy, the investigators also want to propose the optimal dosing guideline of voriconazole with different genetic polymorphisms.

ELIGIBILITY:
Inclusion Criteria: all items below

* male or female ≥ 15 years of age
* immunocompromised patients with hematologic disorders
* patients received voriconazole due to treat proven, probable invasive (pulmonary) aspergillosis

Exclusion Criteria:

* severe hepatic dysfunction (t.bil, AST, ALT, ALP > 5 x upper normal limit)
* who experienced hypersensitivity to azoles
* pregnant women

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematologic malignancies who were given voriconazole to treat invasive (pulmonary) aspergillosis at Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Successful outcome at 12 weeks after voriconazole use | 12 weeks
  Successful outcome = complete response + partial response Unsuccessful outcome = stable disease + failure of therapy + indeterminate response

SECONDARY OUTCOMES:
IFI (invasive fungal infection)-related mortality at 12 weeks | 12 weeks
  IFI (invasive fungal infection)-related mortality at 12 weeks
Successful outcomes at various time points | 1 week, 2 weeks, 4 weeks, and 8 weeks
  Successful outcomes at 1 week,2 weeks,4 weeks, and 8 weeks after voriconazole use
Non-IFI (invasive fungal infection)-related mortality at 12 weeks | 12 weeks
  Non-IFI (invasive fungal infection)-related mortality at 12 weeks
breakthrough IFI | 12 weeks
  breakthrough IFI
Adverse drug reactions | 12 weeks
  Adverse drug reactions (liver function test impairment, visual disturbance, hallucination, photosensitive rash, renal impairment)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea